CLINICAL TRIAL: NCT05660889
Title: Adrenal Vein Sampling as a Tool to Identify Biomarkers That Aid the Diagnosis of Adrenocortical Carcinoma
Acronym: AVS for ACC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Richard Feelders, Principal Investigator, Erasmus Medical Center
Other Study IDs: NL81124.078.22
Record Dates: First submitted 2022-11-24; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Adrenocortical Carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Five patients with strong clinical suspicion of adrenocortical carcinoma
  Interventions: Other: Blood sampling.
- Control group: Twenty patients without suspicion of adrenal malignancy. These patients should undergo an adrenal vein sampling as part of their routine diagnostics.
  Interventions: Other: Blood sampling.

INTERVENTIONS:
Other: Blood sampling. — Blood samples from both study groups, taken during an adrenal vein sampling, will be compared across the groups.

SUMMARY:
The goal of this observational pilot study is to explore whether we can identify biomarkers predictive for the diagnosis of adrenocortical carcinoma in blood. Five participants who are suspected to have adrenocortical carcinoma will undergo an adrenal vein sampling in order to obtain a blood sample from the adrenal vein. This blood sample will be analyzed and compared to blood samples taken from the adrenal vein of 20 control patients, which are patients who do not have adrenocortical carcinoma. The blood samples of the control patients will be drawn during routine medical care.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in the study group, a subject must meet all of the following criteria:

* Patient age ≥18 years
* High clinical suspicion of adrenocortical carcinoma, based on clinical signs (due to hormonal overproduction), steroid hormone profile and radiological features (e.g. tumor size ≥4cm, inhomogenous aspect and tumor attenuation of HU ≥10)
* Able to provide signed informed consent

In order to be eligible to participate in the control group, a subject must meet all of the following criteria:

* Patient age ≥18 years
* Routine diagnostic process includes AVS
* No suspicion of malignancy
* Able to provide signed informed consent

Exclusion Criteria:

Patients are not able to participate if:

* They have a known allergy to (iodinated) contrast fluid
* They use vitamin K antagonizing anticoagulants or DOAC's, except for when on the day of the adrenal vein sampling the anticoagulants are already stopped for the following adrenal surgery, and in case of using vitamin K antagonizing anticoagulants the INR is <3
* The platelet count is below 20
* Anatomy of the adrenal vein is not suitable for performing the AVS procedure, based on the judgement of an experienced interventional radiologist
* Contraindications for use of Synacthen
* They have a known hypersensitivity to any of the substances of Synacthen
* They are pregnant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with a strong clinical suspicion of adrenocortical carcinoma. The control population consists of patients without suspicion of malignancy. The most important for the participants in the control group is that their routine diagnostic tests should include an adrenal vein sampling.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-10-23 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
MicroRNA profile | Analyses will be done at the end of inclusion of all patients, this will be after 2 years. Blood drawn before surgery/treatment will be analysed.
  miRNAs with a log2Fold change > |1| difference in expression in patient compared to control samples.
Presence of mutations in ctDNA | Analyses will be done at the end of inclusion of all patients, this will be after 2 years. Blood drawn before surgery/treatment will be analysed
  Presence of mutations will be assessed in patient samples and compared to control samples
ctDNA methylation pattern | Analyses will be done at the end of inclusion of all patients, this will be after 2 years. Blood drawn before surgery/treatment will be analysed
  Differentially methylated probes and differentially methylated regions will be assessed as those with a beta >0.8 and <0.2
Steroid profile | Analyses will be done at the end of inclusion of all patients, this will be after 2 years. Blood drawn before surgery/treatment will be analysed
  Laboratory values will be compared using Mann-Whitney-U tests

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided